CLINICAL TRIAL: NCT06108466
Title: RELIABILITY AND VALIDITY OF THE DUAL TASK BALANCE TEST IN PATIENTS WITH TOTAL KNEE ARTHROPLASTY
Brief Title: RELIABILITY AND VALIDITY OF THE DT BALANCE TEST IN PATIENTS WITH TKA
Acronym: DT TKA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Ozcan, Msc. Pt, Dokuz Eylul University
Other Study IDs: 6749-GOA
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Knee Injuries and Disorders; Osteo Arthritis Knee
Keywords: Total Knee Arthroplasty; dual test,; timed up and go; reliability
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ability to perform a cognitive task while walking simultaneously is essential in real daily life. However, the psychometric properties of dual-task walking tests have not been well established in patients undergoing total knee arthroplasty (TKA). The aim of study assess the test-retest reliability and validity of dual conditions TUG, 3MBWT, 8FWT nad 4SST in patients with TKA.

ELIGIBILITY:
Inclusion Criteria: TKA -

Exclusion Criteria: revision knee arthroplasty

-

Max Age: 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Total Knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-11-12 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Performance test | 1 Hour
  Timed Up and Go Test
Performance Test | 1 hour
  3MWT
Perfromance Test | 1 hour
  8 FWT
Performance Test | 1 hour
  4SST

OTHER OUTCOMES:
Patient Reported | 1 hour
  HSS Knee Score

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozcan D, Unver B, Karatosun V. Balance assessment under dual task conditions in patients with total knee arthroplasty: a test-retest reliability and concurrent validity study. Physiother Theory Pract. 2025 Jan;41(1):93-98. doi: 10.1080/09593985.2024.2321222. Epub 2024 Feb 21. PMID 38384122